CLINICAL TRIAL: NCT04020770
Title: Influence of Upper Extremity Vibration on Spasticity and Function in Persons With Tetraplegia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shepherd Center, Atlanta GA (Other)
Collaborators: Emory University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Shepherd; FV-765 (Other: Shepherd Center)
Record Dates: First submitted 2019-06-04; First posted 2019-07-16 (Actual); Last update posted 2019-07-16 (Actual); Status verified 2019-07

CONDITIONS: Spinal Cord Injuries; Tetraplegia
MeSH Terms: conditions — Spinal Cord Injuries; Quadriplegia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Vibrating Ball (Experimental): Vibrating ball is held in both hands. Participants complete 5 30-second bouts of 68 Hz vibration with a 1 minute rest in between each bout.
  Interventions: Other: Vibrating ball

INTERVENTIONS:
Other: Vibrating ball — Parameters: 5 30-sec bouts of 68Hz vibration followed by a 1-minute rest.

SUMMARY:
Vibration therapy is a possible alternative to drug-based treatments for spasticity following SCI. Research indicates that it may provide temporary relief from spasticity, but many interventions under investigation are not portable and therefore access is limited. The aim of this study is to investigate the feasibility of using a portable vibrating device to decrease UE spasticity.

ELIGIBILITY:
Inclusion Criteria:

* Have sustained cervical (neurological level C1-C8) SCI
* Any ISNCSCI severity classification (A, B, C or D)
* Have therapist-reported and self-reported spasticity in the arm or hand
* Ability to pick up, move, and release at least one block (on the Box & Blocks Test)
* May participate if utilizing prescription medications, including baclofen pump for control of spasticity

Exclusion Criteria:

* Severe contractures of the arm/hand that limit passive movement of the elbow, wrist or fingers more than 50% of normal range of motion or presence of other orthopedic pathology that would adversely influence participation in the protocol
* Any implanted catheter such as but not limited to CSF shunt, or the presence of pacemaker, implanted automatic internal cardioverter defibrillator (AICD, other cardiac implants and or conditions). Not including baclofen pump.
* Severe pain or hypersensitivity of the arm/hand
* Current pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2018-10-28 (Actual); Primary Completion 2019-02-20 (Actual); Study Completion 2019-02-20 (Actual)

PRIMARY OUTCOMES:
Change in Box and Blocks Test from pre-intervention to post intervention, from pre intervention to 20 minute follow up, from post intervention to 20 minute follow up | Day 1
  Functional assessment of grasp and release
Change in Modified Ashworth Scale from pre-intervention to post intervention, from pre intervention to 20 minute follow up, from post intervention to 20 minute follow up | Day 1
  Clinical assessment of stretch-induced spasticity measured on a scale of 0-4 with 4 indicating the worst spasticity and 0 indicating no spasticity detectable upon clinical examination.
Change in Global Impression of Change Scale from pre-intervention to post intervention, from pre intervention to 20 minute follow up, from post intervention to 20 minute follow up | Day 1
  Self-report of improvement or deterioration over time measured on a scale of 1-7 with 1 indicating very much improved and 7 indicating very much worse
Satisfaction and Adherence Questionnaire | 20 minute delay post intervention
  Self- report of satisfaction with and perceived ability to adhere to the intervention

SECONDARY OUTCOMES:
Hand strength | Pre-intervention, immediately post-intervention, 20 minute delay post intervention
  Dynamometer measurement of grip strength
Pinch strength | Pre-intervention, immediately post-intervention, 20 minute delay post intervention
  Lateral pinch strength measured using a pinch meter
Semmes-Weinstein Monofilament Test | Pre-intervention, immediately post-intervention, 20 minute delay post intervention
  Assesment of light touch sensation
Qualities of Spasticity Questionnaire | Baseline
  Self-report of experience of spasticity

CONTACTS AND LOCATIONS:
Locations (1):
- Shepherd Center, Atlanta, Georgia, United States

IPD SHARING:
Plan to Share IPD: No